CLINICAL TRIAL: NCT06146816
Title: An Exploratory Clinical Trial for the Assessment of Infrared Treatment for Crohn's Disease
Brief Title: The Assessment of Infrared Treatment for Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Sprecher, MD (Other Government)
Responsible Party: Sponsor-Investigator, Eli Sprecher, MD, Professor, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0669-22-TLV
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: IBD; Inflammatory Bowel Diseases; Crohn Disease
Keywords: inflammation; Infra-red
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded, two arms, pilot study. We will recruit 40 CD patients suffering from an active disease based on clinical score and fecal calprotectin level. Thirty patients will be allocated to the experimental group and receive high intensity fIR therapy, while 10 patients will be allocated to the control group and receive the lowest intensity fIR therapy (placebo). Another 10 patients will be recruited in case there is a drop-out. Rate of patients with mild disease (HBI 5-7) will be similar between the two groups.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity fIR therapy (Experimental): Patients will undergo 10 sessions of 30 minutes high intensity fIR therapy at the IBD clinic of the TLVMC by a trained and qualified staff member. Each abdominal quadrant will receive a similar amount of time of exposure to the IR, except for the quadrant of the inflamed intestine (usually the right lower quadrant) which will be exposed longer to the IR. During the treatment, energy levels and skin temperature will be recorded at 10 minutes intervals. Patients responding to therapy (clinical response: ∆HBI≥3 and/or 50% reduction in calprotectin), who did not achieve remission can continue for 10 more treatments.
  Interventions: Device: photobiomodulation treatment in the infrared (IR) range.
- lowest intensity fIR therapy (Placebo Comparator): Patients will undergo 10 sessions of 30 minutes lowest intensity fIR therapy, at the IBD clinic of the TLVMC by a trained and qualified staff member. Each abdominal quadrant will receive a similar amount of time of exposure, except for the quadrant of the inflamed intestine (usually the right lower quadrant) which will be exposed longer. During the treatment, energy levels and skin temperature will be recorded at 10 minutes intervals.
  Interventions: Device: photobiomodulation treatment in the infrared (IR) range.

INTERVENTIONS:
Device: photobiomodulation treatment in the infrared (IR) range. — The baseline treatment included 10 weekly 30 minutes long sessions of fIR treatment.

SUMMARY:
The goal of this clinical trial is to test the safety and efficacy of far Infra-red (fIR) therapy in Crohn's disease patients.

The main questions it aims to answer are:

1. Is infrared therapy safe for treating Crohn's disease patients?
2. Is infrared therapy effective for treating Crohn's disease?

Participants will be asked to attend 10 treatments of fIR therapy, provide stool and blood samples and answer questionnaires.

Researchers will compare between high intensity fIR therapy and lowest intensity fIR therapy (placebo) to see if high intensity fIR therapy is an effective treatment for Crohn's disease.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), are chronic relapsing diseases that carry considerable impact on patients' quality of life, including objective measures such as increased bowel movements, bleeding and fistulas and more subjective measures such as abdominal pain and fatigue.

While the pathogenesis of IBD is thought to result from a deregulated immune response towards microbial antigens in genetically predisposed people, various associations between environmental factors and disease activity have been described. Currently, standard IBD treatment relies on immune modulating drugs. However, such drugs may cause adverse effects, and up to 35% of patients show no response and up to 80% fail to achieve remission.

The investigator would like to explore treating Crohn's disease with photobiomodulation in the infrared (IR) range. Preliminary data suggest a positive effect of IR on Crohn's disease activity, and would like to conduct a small scale, pilot clinical trial to further clinically explore the safety and efficacy of this simple intervention.

Infrared is a safe, non-ionizing radiation spanning wavelengths from about 800 nanometers (nm) to 1 millimeter (mm). The therapeutic effects of IR radiation were serendipitously stumbled upon in the 1980s by NASA (National Aeronautics and Space Administration) scientists who noticed improvement in skin lesions when assessing IR light for growing potatoes in space. Since then, there has been a cautious advancement in assessing IR therapy for various conditions and an increased understanding of some of the mechanisms underlying its effect.

Alongside its beneficial effect, infrared treatment is not associated with serious adverse effects in general and with relation to fertility in particular. In fact, experimental data suggest that far IR (fIR) is safe for treating various medical conditions including cancer, diabetes and female infertility.

Due to the documented effects of IR therapy on inflammation and its favorable safety profile, the investigator would like to assess its effect on Crohn's disease. A skilled staff member will use a device emitting fIR radiation (8-10 microns) that is able to penetrate deep into the body (up to at least 20 cm according to manufacturer). The device comprises a heating pad that emits heat (up to 70 degree C) alongside fIR radiation.

Prior to treatment patient's bowel will be assessed by intestinal ultrasound (IUS) / CT/ MRI to determine the location of inflammation in order to focalize treatment, but also to rule out the presence of abscess and cysts.

All patients will undergo 10 sessions of 30 minutes fIR therapy at the IBD clinic of the Tel Aviv Medical Center (TLVMC) by a trained and qualified staff member. Each abdominal quadrant will receive a similar amount of time of exposure to the IR, except for the quadrant of the inflamed intestine (usually the right lower quadrant) which will be exposed longer to the IR. During the treatment, energy levels and skin temperature will be recorded at 10 minutes intervals.

Patients responding to therapy (clinical response: ∆HBI≥3 and/or 50% reduction in calprotectin), who did not achieve remission can continue for 10 more treatments. Patients who are allocated to the control group will be eligible to transfer to the experimental group after 10 sessions and receive 10 treatments with a high intensity fIR.

After the completion of treatments, at week 11, bowel thickness will be assessed again by IUS, as well as biochemical and clinical indexes.

Clinical score will be assessed using the Harvey-Bradshaw index (HBI) at weeks: 0, 5, and 10.

Stool will be collected at weeks 0, 5 and 10 for fecal calprotectin analysis and for future microbiome/proteomics analysis.

Blood will be collected at weeks 0, 5, and 10 for C reactive protein (CRP), complete blood count (CBC), liver function tests, creatinine and lipase. Serum will be frozen for future proteomics and inflammatory measures analysis. Total blood volume will be less than 20ml.

Patients will be asked to complete questionnaires evaluating their quality of life and disease related symptoms and outcomes.

Side effects such as local skin thermal injury and blood tests abnormalities will be documented. In case of local skin thermal injury, patients will be examined to determine injury level, with recommendation to apply Aloe Vera paste and a follow-up call will be made to document resolution of symptoms within 2 days.

Throughout the research period patients will be asked to maintain their usual lifestyle with regards to nutrition and physical activity habits

Statistics Test results, clinical indexes and side effects will be compared between experimental and control groups prior to- and post treatment. These measures will also be analyzed within groups to compare pre- and post-treatment results.

Patients in both groups will be categorized by disease severity level (according to HBI) in order to correlate disease severity with treatment efficacy. Patients will be randomized according to disease severity in order to keep an equal rate of patients with mild clinical disease activity upon recruitment.

All statistical analyses will be performed using SPSS version 23.0 for Windows. Demographic characteristics of the population will be described by mean±SD for continuous variables, while categorical variables will be displayed as a frequency table.

Normal distribution will be tested by Kolmogorov-Smirnov test. If normality is rejected, non-parametric tests will be used.

ELIGIBILITY:
Inclusion Criteria:

1. An established Crohn's disease
2. 18 < age < 80
3. No therapy or on constant medicinal regimen throughout the study period: mesalamine at least 6 weeks, or steroids at least 2 weeks, or immunomodulatory drugs at least 12 weeks or biologics at least 12 weeks, medical cannabis at least 2 weeks before the study.
4. CD patients will be included if their symptoms score >4 on the Harvey-Bradshaw index (HBI) score and/or fecal calprotectin level > 150 ug/gr.

Exclusion Criteria:

1. BMI greater than 30 Kg/m2
2. Any proven current infection such as Clostridioides difficile infection, positive stool culture, or parasites.
3. Inability to sign informed consent and complete study protocol
4. Pregnancy
5. Subjects with chronic conditions such as cancer, organ transplant subjects, advanced kidney or liver disease, systemic inflammatory conditions other than IBD.
6. Presence of abscess and cysts in the liver/ kidneys or pancreas
7. Evidence of an abdominal abscess or entero-enteric fistula.
8. More than one CD luminal surgery or a small bowel length < 1.5 meter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of fIR therapy for CD patients. | 2 years
  We will document all adverse events and assess their severity. The only documented adverse event for fIR treatment in the currently available literature are first degree burns. Hence, the treatment will be considered safe if we will not encounter additional adverse events. Clinical and biochemical markers will be monitored for the possibility of disease exacerbation following fIR treatment.

SECONDARY OUTCOMES:
Assess the efficacy of high intensity fIR compared to low intensity fIR in achieving a composite response. | 3 years
  a composite response rate defined as a clinical response (drop of ≥3 points of the Harvey-Bradshaw Index (HBI) or HBI<5) AND a decrease of fecal calprotectin (Fcal) by at least 50% from baseline or Fcal<150ug/gr.
Assess the efficacy of high intensity fIR compared to low intensity fIR in achieving Clinical remission. | 3 years
  Clinical remission is defined by HBI≤4
Assess the efficacy of high intensity fIR compared to low intensity fIR in achieving biomarker remission. | 3 years
  Biomarker remission is defined by normalization of Fcal<150ugr/g
Assess the efficacy of high intensity fIR compared to low intensity fIR by rate of sonographic healing. | 3 years
  Measure rate of sonographic healing as assessed by IUS (intestinal ultrasound) and defined as bowel wall thickening ≤3 mm with no increase in color Doppler signal.

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, Professor, Principal Investigator — Department of Gastroenterology and Liver Diseases, Tel Aviv Medical Center, Tel Aviv, Israel
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No